CLINICAL TRIAL: NCT06517069
Title: Effect of Transcutaneous Electrical Acupoint Stimulation Combined With Oxycodone on Postoperative Visceral Pain and Early Recovery Quality in Gynecologic Laparoscopic Patients
Brief Title: Effect of TEAS Combined With Oxycodone on Postoperative Visceral Pain in Gynecologic Laparoscopic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Wang wanxia, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kang
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Visceral Pain
MeSH Terms: conditions — Visceral Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TEAS combined with Oxycodone (Experimental): Bilateral Neiguan point (PC6), Zusanli point (ST36) and Sanyinjiao point (SP6) were selected. Use Huatuo electronic needle therapy device, Sulodine electric stimulation hand circle TEAS, Huatuo electronic needle therapy device parameter setting: Density wave, 2/10Hz, current intensity from weak to strong, until the patient can tolerate the maximum intensity (acid, numbness, distension, pain) is appropriate, after the Sulodine brand electrical stimulation bracelet is turned on, gradually increase the stimulation intensity, until the patient can tolerate the maximum intensity is appropriate, stimulation for 30min until anesthesia induction; Oxycodone 0.1mg/kg was injected intravenously 5 minutes before anesthesia induction
  Interventions: Other: TEAS; Drug: Oxycodone
- TEAS (Experimental): Bilateral Neiguan point (PC6), Zusanli point (ST36) and Sanyinjiao point (SP6) were selected. Use Huatuo electronic needle therapy device, Sulodine electric stimulation hand circle TEAS, Huatuo electronic needle therapy device parameter setting: Density wave, 2/10Hz, current intensity from weak to strong, until the patient can tolerate the maximum intensity (acid, numbness, distension, pain) is appropriate, after the Sulodine brand electrical stimulation bracelet is turned on, gradually increase the stimulation intensity, until the patient can tolerate the maximum intensity is appropriate, stimulation for 30min until anesthesia induction; The same amount of normal saline was injected intravenously 5 minutes before anesthesia induction.
  Interventions: Other: TEAS
- Oxycodone (Experimental): Bilateral Neiguan point (PC6), Zusanli point (ST36) and Sanyinjiao point (SP6) were selected. Stick electrodes only but do not stimulate; Oxycodone 0.1mg/kg was injected intravenously 5 minutes before anesthesia induction
  Interventions: Drug: Oxycodone
- Comparator (No Intervention): Bilateral Neiguan point (PC6), Zusanli point (ST36) and Sanyinjiao point (SP6) were selected. Stick electrodes only but do not stimulate; The same amount of normal saline was injected intravenously 5 minutes before anesthesia induction.

INTERVENTIONS:
Other: TEAS — Bilateral Neiguan point (PC6), Zusanli point (ST36) and Sanyinjiao point (SP6) were selected. Use Huatuo electronic needle therapy device, Sulodine electric stimulation hand circle TEAS, Huatuo electronic needle therapy device parameter setting: Density wave, 2/10Hz, current intensity from weak to strong, until the patient can tolerate the maximum intensity (acid, numbness, distension, pain) is appropriate, after the Sulodine brand electrical stimulation bracelet is turned on, gradually increase the stimulation intensity, until the patient can tolerate the maximum intensity is appropriate, stimulation for 30min until anesthesia induction
  Arms: TEAS; TEAS combined with Oxycodone
Drug: Oxycodone — Oxycodone 0.1mg/kg was injected intravenously 5 minutes before anesthesia induction
  Arms: Oxycodone; TEAS combined with Oxycodone

SUMMARY:
To investigate the effect and feasibility of percutaneous acupoint stimulation combined with oxycodone on postoperative visceral pain in laparoscopic patients, and provided a clinical basis for optimizing perioperative pain management in laparoscopic patients.

DETAILED DESCRIPTION:
Patients aged 18-65 years old, BMI 18-30kg/m2, ASA grade I or II were selected for gynecologic laparoscopic surgery (laparoscopic ovarian tumor stripping, laparoscopic uterine fibroid stripping, laparoscopic total hysterectomy) under general anesthesia from May 2024 to July 2024. Exclusion criteria: Patients who were allergic to the drugs used in the study, had confusion or cognitive impairment, contraindicated percutaneous acupoint electrical stimulation, abnormal cardiopulmonary and liver and kidney function, history of analgesic drug use within one week, history of diabetes, myocardial infarction, or cerebrovascular accident. Exclusion criteria: patients dropped out of the experiment midway or the data was not completely collected, the surgical method changed midway, the operation duration was less than 30 minutes or more than 2 hours, and patients with opioid and addictive drug dependence

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* American Society of Anesthesiologists grade I-II
* Body mass index (BMI) 18.5-30 kg/m2;
* No ulceration or infection at the acupuncture stimulation site.

Exclusion Criteria:

* Allergic to the drugs used in the study;
* People with unclear consciousness or cognitive dysfunction;
* There are contraindications of percutaneous acupoint electrical stimulation;
* Abnormal cardiopulmonary and liver and kidney function;
* History of analgesic drug use within one week;
* History of diabetes, myocardial infarction or cerebrovascular accident.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
the VAS score of postoperative visceral pain | 30 minutes after surgery、6 hours after surgery、24 hours after surgery、48 hours after surgery
  the visual analogue scale of postoperative visceral pain,The basic method is to use a swimming scale about 10cm long, marked with 10 scales on one side, and "0" and "10" at each end, with 0 being painless and 10 being the most unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China